CLINICAL TRIAL: NCT06044272
Title: Antimicrobial Resistance Profiles in Healthcare Facilities From Meta State, Colombia: A Retrospective Observational Study From 2018-2022
Brief Title: Antimicrobial Resistance in Hospitals From Meta, Colombia
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, Principal investigator, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2023_03_RAM
Record Dates: First submitted 2023-07-20; First posted 2023-09-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Increased Drug Resistance
Keywords: Patient Safety; Healthcare Quality Assurance; Cross Infection; Increased Drug Resistance; Colombia
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Escherichia coli producing ESBL: Ceftazidime or cefotaxime resistance.
  Interventions: Other: Factors associated
- Klebsiella pneumoniae producing ESBL: Ceftazidime or cefotaxime resistance.
  Interventions: Other: Factors associated
- Klebsiella pneumoniae resistant to carbapenem: Ertapenem resistance.
  Interventions: Other: Factors associated
- Pseudomonas aeruginosa resistant to carbapenems: Imipenem or meropenem resistance.
  Interventions: Other: Factors associated
- Staphylococcus aureus resistant to methicillin: Methicillin resistance.
  Interventions: Other: Factors associated

INTERVENTIONS:
Other: Factors associated — Factors associated with the type of resistance by microorganisms.

SUMMARY:
Introduction: Healthcare-associated infections cause a burden in morbidity and mortality, and they increase the financial cost of care. Nevertheless, they are not limited to setting factors, and several community conditions and contexts are linked. Clinical laboratories from hospitals report monthly to the Public Health Laboratory.

Objective: The study aims to establish the antimicrobial resistance profile of the most significant bacteria involved in healthcare-associated infections in Meta State hospitals.

Methodology: The researchers designed a retrospective observational trial with the records from samples and origin, microbial findings, and antibiogram. The outcome was the mechanism for antimicrobial resistance. The information from the State Public Health Laboratory database was exported to Excel for analysis.

Conclusions: The outlook of Enterobacteriaceae and Staphylococcus aureus antimicrobial resistance in hospitals from Meta State will be revealed. Comprehensive strategies for mitigation, including continuous microbiological surveillance, are needed.

DETAILED DESCRIPTION:
Healthcare-associated infections (HCAIs) affect patients' security and quality of care. Several of them develop infections during their hospital stay, especially in the ICU, and the number is higher in low-middle-income countries. It confers an additional burden on hospitals, with higher use of resources and costs. The magnitude of the problem is not understood completely due to discrepancies in results and heterogeneous studies.

Additionally, HCAIs are associated with increased morbidity and disability, but the studies are unsure of the effect on mortality.

Microorganisms are ubiquitous in hospital environments and diverse in patients, families, and healthcare personnel. Some are carriers of antimicrobial resistance mechanisms (AMR) and are transmissible to other microorganisms. Studies with genetic sequencing show a fundamental role of such colonization as a reservoir for AMR that limits the efficacy of therapy since admission. Such technology is not available to most hospitals to screen environments or people. Such interaction favors an interchange of microbiome (directly or indirectly) as a requirement for the advent of HCAIs.

It is known that HCAIs by MDR (multidrug resistance) bacteria are associated with an increase in mortality (OR 1.61; 1.36-1.90); it is not clear if it is due to the problem in the quality of care or the health conditions that promotes the infection.

The frequency of HCAIs is higher in Latin America than in the United States or Europe. The Centers for Disease Control and Prevention regularly monitor DAI (device-associated infections) from several years ago, and they are of reference worldwide.

Some countries have developed microbiological surveillance systems to follow up on changes in resistance phenotypes. They reveal benign resistance patterns in Gram-negative in contrast to the reports from studies in Colombia. Such results highlight the importance of analyzing the information provided by such monitoring to prioritize actions and resources to modulate the impact of the increased resistance.

ELIGIBILITY:
Inclusion Criteria:

* All records with results from microbial isolation and antimicrobial resistance profile.

Exclusion Criteria:

* Records of quality control; no information on resistance or susceptibility.

Max Age: 130 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population included in the study were the records of microbiological isolation for surveillance from the Public Health Laboratory of Meta State Secretary of Health.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of microorganisms resistant to the antimicrobial | 28 days
  Mechanism of resistance by type of microorganisms. ESBL in E. coli and K. pneumoniae, carbapenemase in K.pneumoniae and Pseudomonas, and methicilinase in S. aureus.

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Cooperative University of Colombia
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The database is access restricted in the university repository.

REFERENCES:
- [Result] Kawata S, Morimoto S, Kosai K, Kawamoto Y, Nakashima Y, Morinaga Y, Yanagihara K, Yoshida LM, Moriuchi H. The fecal carriage rate of extended-spectrum beta-lactamase-producing or carbapenem-resistant Enterobacterales among Japanese infants in the community at the 4-month health examination in a rural city. Front Cell Infect Microbiol. 2023 Jun 14;13:1168451. doi: 10.3389/fcimb.2023.1168451. eCollection 2023. PMID 37389210
- [Result] Zhou Y, Zhou S, Peng J, Min L, Chen Q, Ke J. Bacterial distribution and drug resistance in blood samples of children in Jiangxi Region, 2017-2021. Front Cell Infect Microbiol. 2023 Jun 22;13:1163312. doi: 10.3389/fcimb.2023.1163312. eCollection 2023. PMID 37424793
- [Result] Quiros RE, Bardossy AC, Angeleri P, Zurita J, Aleman Espinoza WR, Carneiro M, Guerra S, Medina J, Castaneda Luquerna X, Guerra A, Vega S, Cuellar Ponce de Leon LE, Munita J, Escobar ED, Maki G, Prentiss T, Zervos M; PROA-LATAM Project Group. Antimicrobial stewardship programs in adult intensive care units in Latin America: Implementation, assessments, and impact on outcomes. Infect Control Hosp Epidemiol. 2022 Feb;43(2):181-190. doi: 10.1017/ice.2021.80. Epub 2021 Apr 8. PMID 33829982
- [Result] Sharma A, Luvsansharav UO, Paul P, Lutgring JD, Call DR, Omulo S, Laserson K, Araos R, Munita JM, Verani J, Chowdhury F, Muneer SM, Espinosa-Bode A, Ramay B, Cordon-Rosales C, Kumar CPG, Bhatnagar T, Gupta N, Park B, Smith RM. Multi-country cross-sectional study of colonization with multidrug-resistant organisms: protocol and methods for the Antibiotic Resistance in Communities and Hospitals (ARCH) studies. BMC Public Health. 2021 Jul 16;21(1):1412. doi: 10.1186/s12889-021-11451-y. PMID 34271883
- [Result] Alzamora MC, Echevarria AC, Ferraro VM, Riveros MD, Zambruni M, Ochoa TJ. [Antimicrobial resistance of commensal Escherichia coli strains in children of two rural communities in Peru]. Rev Peru Med Exp Salud Publica. 2019 Jul-Sep;36(3):459-463. doi: 10.17843/rpmesp.2019.363.4366. Epub 2019 Dec 2. Spanish. PMID 31800939
- [Result] Revoredo Rego F, Huaman Egoavil E, Zegarra Cavani S, Auris Mora H, Valderrama Barrientos R. [Microbiological and resistance profiles of community acquired and nosocomial intra abdominal infections in surgery of National Hospital Guillermo Almenara, Lima, Peru]. Rev Gastroenterol Peru. 2016 Apr-Jun;36(2):115-22. Spanish. PMID 27409087
- [Result] Vallejo M, Cuesta DP, Florez LE, Correa A, Llanos CE, Isaza B, Vanegas S, Osorio J, Casanova L, Villegas MV. [Clinical and microbiological characteristics of complicated intra-abdominal infection in Colombia: a multicenter study]. Rev Chilena Infectol. 2016 Jun;33(3):261-7. doi: 10.4067/S0716-10182016000300002. Spanish. PMID 27598273
- [Result] Arias-Flores R, Rosado-Quiab U, Vargas-Valerio A, Grajales-Muniz C. [Microorganisms responsible of nosocomial infections in the Mexican Social Security Institute]. Rev Med Inst Mex Seguro Soc. 2016 Jan-Feb;54(1):20-4. Spanish. PMID 26820194
- [Result] Mata-Hernandez A, Rivera-Villa AH, Miguel-Perez A, Perez-Atanasio JM, Torres-Gonzalez R. [Sensitivity and antibiotic resistance in infections of the musculoskeletal system]. Rev Med Inst Mex Seguro Soc. 2016;54 Suppl 3:S320-S324. Spanish. PMID 27855057
- [Result] Morganti L, Cordova E, Cassini E, Gomez N, Lopez Moral L, Badia M, Rodriguez C. [Antimicrobial susceptibility of Gram-negative bacilli of community acquired intra-abdominal infections in a hospital at Buenos Aires, Argentina]. Rev Esp Quimioter. 2016 Aug;29(4):202-5. Epub 2016 Jun 17. Spanish. PMID 27318458
- [Result] Ruiz-Garbajosa P, Canton R. [Epidemiology of multi-drug resistant gramnegative bacilli]. Rev Esp Quimioter. 2016 Sep;29 Suppl 1:21-5. Spanish. PMID 27608308
- [Result] De La Rosa G, Leon AL, Jaimes F. [Epidemiology and prognosis of patients with bloodstream infection in 10 hospitals in Colombia]. Rev Chilena Infectol. 2016 Apr;33(2):141-9. doi: 10.4067/S0716-10182016000200003. Spanish. PMID 27314991
- [Result] Salgado P, Gilsanz F, Maseda E. [Resistant gram-negative bacteria. Therapeutic approach and risk factors]. Rev Esp Quimioter. 2016 Sep;29 Suppl 1:26-30. Spanish. PMID 27608309
- [Result] Moya-Dionisio V, Diaz-Zabala M, Ibanez-Fernandez A, Suarez-Leiva P, Martinez-Suarez V, Ordonez-Alvarez FA, Santos-Rodriguez F. [Uropathogen pattern and antimicrobial susceptibility in positive urinary cultures isolates from paediatric patients]. Rev Esp Quimioter. 2016 Jun;29(3):146-50. Epub 2016 Apr 19. Spanish. PMID 27092771
- [Result] Cercenado E. [Epidemiology of the infection by resistant Gram-positive microorganisms]. Rev Esp Quimioter. 2016 Sep;29 Suppl 1:6-9. Spanish. PMID 27608305
- [Result] Cercenado E. [Laboratory detection of carbapenemase-producing Enterobacteriaceae]. Rev Esp Quimioter. 2015 Sep;28 Suppl 1:8-11. Spanish. PMID 26365726
- [Result] Betran A, Cortes AM, Lopez C. [Evaluation of antibiotic resistance of Escherichia coli in urinary tract infections in Primary Care Barbastro Sector (Huesca)]. Rev Esp Quimioter. 2015 Oct;28(5):263-6. Spanish. PMID 26437757
- [Result] Gutiérrez Lesmes OA. [Resistance and susceptibility of microorganisms isolatedin patients treated in a tertiary institution hospital, Villavicencio-Colombia, 2012]. Rev Cuid. 2015 May 15;6(1):947-54.
- [Result] Ocampo AM, Vargas CA, Sierra PM, Cienfuegos AV, Jimenez JN. [Molecular characterization of an outbreak of carbapenem-resistant Klebsiella pneumoniae in a tertiary care hospital in Medellin, Colombia]. Biomedica. 2015 Oct-Dec;35(4):496-504. doi: 10.7705/biomedica.v35i4.2610. Spanish. PMID 26844438
- [Result] Pérez N, Pavas N, Rodríguez EI. Resistencia a los antibióticos en Escherichia coli con beta-lactamasas de espectro extendido en un hospital de la Orinoquia colombiana. Infectio. 2011;15(3):147-54.